CLINICAL TRIAL: NCT05922332
Title: Application and Effect Evaluation of Medium Chain Fatty Acid Rich Milk Powder in Infants With Cholestatic Liver Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study could not be conducted as a randomized controlled study due to a change in the protocol, and the study needs to be stopped.
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHFudanU0530
Record Dates: First submitted 2023-06-04; First posted 2023-06-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cholestatic Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rich medium chain fatty acid milk powder group (Experimental): This group will be fed milk powder rich in medium-chain fatty acids. The MCT content of formula milk is 39%, and the total energy is 68kcal/100ml.
  Interventions: Dietary Supplement: Rich medium chain fatty acid milk powder group
- Regular milk powder group (Active Comparator): This group will be fed regular milk powder.The MCT content of formula milk is less than 30%, and the total energy is 67kcal/100ml.
  Interventions: Dietary Supplement: Regular milk powder group

INTERVENTIONS:
Dietary Supplement: Rich medium chain fatty acid milk powder group — In intervention group,there are 32 infants.They will be fed with rich medium chain fatty acid milk powder, formula with MCT content of 39%, total energy of 68kcal/100ml, and feeding frequency at a 3-hour interval
  Arms: Rich medium chain fatty acid milk powder group
Dietary Supplement: Regular milk powder group — In control group,there are 32 infants.They will be fed regular milk powder,formula with MCT content of less than 30%, total energy of 67kcal/100ml, and feeding frequency at a 3 hours interval
  Arms: Regular milk powder group

SUMMARY:
To verify the effect of feeding milk powder rich in medium chain fatty acids on improving the nutritional status and disease status of infants with cholestatic liver disease and To evaluate the safety of feeding milk powder rich in medium chain fatty acids in infants with cholestatic liver disease.

DETAILED DESCRIPTION:
This study will include all types of cholestatic liver disease in infants, randomized controlled study of the efficacy and safety of intervention with rich medium chain fatty acid milk powder,To verify the effect of feeding milk powder rich in medium chain fatty acids on improving the nutritional status and disease status of infants with cholestatic liver disease .

ELIGIBILITY:
Inclusion Criteria:

* meets the diagnostic criteria of cholestasis
* Artificial feeding (formula feeders)
* Age ≤6 months
* The course of cholestasis was > 1 month
* Informed consent of the guardian

Exclusion Criteria:

* There are major non-cholestatic genetic diseases leading to nutritional intake disorders, such as gastrointestinal malformations
* Cholestasis with ascites and diarrhea
* In patients with oxidative impairment of medium chain fatty acids

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Z-scores of weight for age | "from enrollment to the 4 weekend(28 days)"
  The change of WAZ would be calculation at the 4 weekend(28 days) after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Children's Hospital of Fudan University Children's Hospital of Fudan University, Study Chair — employee
Locations (1):
- zhaoyang Gou, Shanghai, China

IPD SHARING:
Plan to Share IPD: No